CLINICAL TRIAL: NCT06699446
Title: The "Seamless" Patient: From Preoperative Preparation to Postoperative Rehabilitation
Brief Title: The "Seamless" Patient:From Preoperative Preparation to Postoperative Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01VSF21036
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care" (No Intervention): Previous postal call-in without additional communication or special follow-up
- Intensified patient education (Other): via classical communication channels as well as provision of information material for outpatient, preoperative pre-rehabilitation (respiratory training, exercise therapy). Establish an individualized rehabilitation plan and telephone postoperative communication (postoperative for Patient-Reported Experience Measures (PREMs) and Patient-Reported Outcome Measures (PROM) analysis) with the surgical center
  Interventions: Other: pre rehabilitation
- Intensified education on new media (mobile app) (Other): with outpatient preoperative rehabilitation (respiratory training, exercise therapy). Creation of an individualized rehabilitation plan and postoperative, two-way communication via mobileapp.
  Interventions: Other: pre rehabilitation

INTERVENTIONS:
Other: pre rehabilitation — preoperative pre-rehabilitation (respiratory training, exercise therapy). Establish an individualized rehabilitation plan and postoperative communication via telephone or app
  Arms: Intensified education on new media (mobile app); Intensified patient education

SUMMARY:
The "seamless" patient: from preoperative preparation to postoperative rehabilitation.

The effects of digital services for perioperative care of patients undergoing cardiac surgery will be investigated

DETAILED DESCRIPTION:
Intervention by randomization in: G1. "Standard of care" Previous postal call-in without additional communication or special follow-up G2: Intensified patient education via classical communication channels as well as provision of information material for outpatient, preoperative pre-rehabilitation (respiratory training, exercise therapy). Establish an individualized rehabilitation plan and telephone postoperative communication (postoperative for Patient-Reported Experience Measures (PREMs) and Patient-Reported Outcome Measures (PROM) analysis) with the surgical center. G3: Intensified education on new media (mobile app) with outpatient preoperative rehabilitation (respiratory training, exercise therapy). Creation of an individualized rehabilitation plan and postoperative, two-way communication via mobileapp.

This project combines the establishment of outpatient pre-rehabilitation with the additional benefit of interrogating patient-reported outcome (PROs) with individualized rehabilitation. Through the improved exchange of information and the resulting more intensive care of patients alone, we hope not only to improve the quality of life, but also to reduce postoperative mortality and morbidity. The use of new techniques with the establishment of a mobile-based app should provide a decisive advantage in the effectiveness of the measures in this regard. The integration of secure, direct, and always-available communication channels will both improve the flow of information and enhance patients' sense of security in an increasingly fast-moving healthcare system.

Hypotheses:

* The intervention in G2 "classic forms of communication" does not significantly improve the primary and secondary endpoints compared to the control group G1.
* The intervention in G3 "next level" communication via app leads to a significant improvement of the primary and secondary endpoints compared to control group G1.
* The rate of exercise performance (in the prehabilitation and rehabilitation phases; % of days) is significantly higher in the G3 "next level" communication via app group compared to the G2 "classical forms of communication" group.
* Intervention in G2 "classical forms of communication" and G3 "next level" communication via app leads to significant improvement in PREMs compared to control group G1.
* The questionaires: EQ-VAS, PROMIS-10 and HSSI are equally suitable for mapping the health status of patients* in the postoperative course.
* The feedback rate (completion of the query) on health status is significantly higher for the questionaires EQ-VAS compared to questionaire PROMIS-10, questionaire HSSI and questionaire MLHFQ.
* In patients* who develop postoperative pericardial tamponade, pneumonia, or surgical access wound complication (bleeding/Dressler syndrome, infection/sepsis, wound dehiscence/infection, mechanical instability), Questionaire EQ-VAS scores drop significantly before diagnosis. The questionaire EQ-VAS is therefore suitable as a non-specific postoperative parameter for triggering early further diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Patient is capable of giving consent;
* planned, elective cardiac surgery (coronary bypass surgery and heart valve surgery incl. combination surgery). The planned surgery can be performed with or without a heart-lung machine.
* Minimally invasive procedures may also be explicitly included in the study.

Exclusion Criteria:

* Emergency care;
* congenital heart defects;
* age less than 18 years;
* patient unable to give consent;
* patient unable to perform simple physical training;
* high-risk surgery with a calculated Euroscore II of more than 8%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life of patient via questionnaire | 6 month
  via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School Hanover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No